CLINICAL TRIAL: NCT00120224
Title: De-Medicalizing Mifepristone Medical Abortion
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Collaborators: Planned Parenthood Federation of America (Other); David and Lucile Packard Foundation (Other)
Other Study IDs: 1.1.2
Record Dates: First submitted 2005-06-30; First posted 2005-07-15 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Medical Abortion
Keywords: Mifepristone; Medical abortion; Ultrasound

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This study will investigate the possibility that medical abortion using mifepristone and misoprostol - a safe, proven therapy for terminating early first trimester pregnancy - can be administered in a manner that is simpler and less costly than that routinely employed in the United States.

The researchers hypothesize that:

1. Practitioners themselves, based on history and examination but without sonography, are able to dependably and correctly determine which patients are eligible for medical abortion and which patients either are not eligible or require further evaluation to determine eligibility.
2. Practitioners themselves, based on a symptom diary and low-sensitivity pregnancy test but without sonography, are able to dependably and correctly determine when a successful medical abortion has taken place and when referral for other possible outcomes should be made.
3. A symptom diary and low-sensitivity pregnancy test are safe and effective means of separating those women who could benefit from a follow-up visit from those who do not need one.

DETAILED DESCRIPTION:
Mifepristone medical abortion has been available in France for a decade and a half and in the United States since 2001. Over this time, it has been demonstrated to be as safe as or safer than either surgical abortion or carrying a pregnancy to term. Furthermore, as medical abortion employs medications rather than surgery to terminate a pregnancy, it has the potential to greatly increase the availability of locations providing abortion services in the US, eliminating as it does the need for expensive equipment and surgical training.

Unfortunately, however, although the availability of medical abortion in the US has increased with time, it has yet to achieve its full potential. In large part this appears to be due to two factors which inhibit providers from offering, and women from choosing, the procedure: 1) Although the approved US medical abortion regimen does not require providers to use ultrasound examination as part of the procedure, it has become common practice for providers to do so. This both increases the cost of the procedure and limits the number of facilities that can offer it. 2) While surgical abortion typically requires only one clinic visit, medical abortion requires (officially) three or (in practice) two visits, making it more expensive, less convenient, and less attractive to women.

There is already a great deal of evidence that medical abortion can be safely offered with two (or even fewer) office visits, and without routine ultrasonography. Most medical abortions in the United States, in fact, currently require only two visits, and the possibility exists that women could self-screen at home, based on a symptom checklist, to determine if the second of these (the follow-up visit) is necessary - an approach that could spare the large majority of medical abortion clients who have uncomplicated courses an extra trip to the clinic. There are, in addition, several less-expensive and less technology-intensive approaches to gathering the diagnostic information currently being provided, pre- and post-procedure, by ultrasonography.

The purpose of the current study is to test the feasibility and efficacy of an approach to medical abortion that forgoes the routine use of ultrasonography. It will also provide evidence on the feasibility of eliminating the requirement for a universal follow-up visit based on self-screening by medical abortion clients. In providing data to make these tests, however, the study protocol will not in any way abridge the medical abortion care currently received by clients at the participating facilities. The study will permit clients to receive standard care (including a follow-up visit and pre- and post-procedure ultrasound examinations in all cases) while gathering valuable information which, we hope, will provide a basis for simplifying standard care in the future.

The research questions to be answered by the study are:

1. Do an interview with the abortion client, a pregnancy test and a physical exam provide adequate information to determine which abortion clients are eligible for the medical abortion procedure and which should be referred for sonography (or other diagnostic tests) before making such a determination?
2. Can a self-administered symptom diary and a follow-up low-sensitivity pregnancy test provide an adequate basis to determine whether a woman has undergone a successful medical abortion or whether she requires a sonographic exam (or other diagnostic test) in order to make this determination?
3. Does a post-abortion pelvic examination provide valuable additional information for determining whether a woman has undergone a successful medical abortion or whether she requires a sonographic exam (or other diagnostic test) in order to make this determination?
4. Can a self-administered symptom diary and a low-sensitivity pregnancy test provide an adequate basis for determining which medical abortion clients require a follow-up visit?

The research hypotheses are:

1. Practitioners themselves, based on history and examination but without sonography, are able to dependably and correctly determine which patients are eligible for medical abortion and which patients either are not eligible or require further evaluation to determine eligibility.
2. Practitioners themselves, based on a symptom diary and low-sensitivity pregnancy test but without sonography, are able to dependably and correctly determine when a successful medical abortion has taken place and when referral for other possible outcomes should be made.
3. A symptom diary and low-sensitivity pregnancy test are safe and effective means of separating those women who could benefit from a follow-up visit from those who do not need one.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting at study clinics for medical abortion who agree to complete home study card and return for follow-up visit

Exclusion Criteria:

* Women presenting at study clinics for medical abortion who do not agree to participate in study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4410
Dates: Start 2005-05; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Clark, MPH, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (3):
- United States (3):
  - Planned Parenthood of San Diego and Riverside Counties, San Diego, California
  - Family Planning Associates Medical Group, Chicago, Illinois
  - Planned Parenthood of New York City, New York, New York

REFERENCES:
- [Background] Savitz DA, Terry JW Jr, Dole N, Thorp JM Jr, Siega-Riz AM, Herring AH. Comparison of pregnancy dating by last menstrual period, ultrasound scanning, and their combination. Am J Obstet Gynecol. 2002 Dec;187(6):1660-6. doi: 10.1067/mob.2002.127601. PMID 12501080
- [Background] Taipale P, Hiilesmaa V. Predicting delivery date by ultrasound and last menstrual period in early gestation. Obstet Gynecol. 2001 Feb;97(2):189-94. doi: 10.1016/s0029-7844(00)01131-5. PMID 11165580
- [Background] Mongelli M, Wilcox M, Gardosi J. Estimating the date of confinement: ultrasonographic biometry versus certain menstrual dates. Am J Obstet Gynecol. 1996 Jan;174(1 Pt 1):278-81. doi: 10.1016/s0002-9378(96)70408-8. PMID 8572021
- [Background] Fielding SL, Schaff EA, Nam NY. Clinicians' perception of sonogram indication for mifepristone abortion up to 63 days. Contraception. 2002 Jul;66(1):27-31. doi: 10.1016/s0010-7824(02)00316-5. PMID 12169378
- [Background] Barnhart KT, Simhan H, Kamelle SA. Diagnostic accuracy of ultrasound above and below the beta-hCG discriminatory zone. Obstet Gynecol. 1999 Oct;94(4):583-7. doi: 10.1016/s0029-7844(99)00347-6. PMID 10511363
- [Background] Fiala C, Safar P, Bygdeman M, Gemzell-Danielsson K. Verifying the effectiveness of medical abortion; ultrasound versus hCG testing. Eur J Obstet Gynecol Reprod Biol. 2003 Aug 15;109(2):190-5. doi: 10.1016/s0301-2115(03)00012-5. PMID 12860340
- [Derived] Clark W, Bracken H, Tanenhaus J, Schweikert S, Lichtenberg ES, Winikoff B. Alternatives to a routine follow-up visit for early medical abortion. Obstet Gynecol. 2010 Feb;115(2 Pt 1):264-272. doi: 10.1097/AOG.0b013e3181c996f3. PMID 20093898
- See also: Related Info — http://www.gynuity.org